CLINICAL TRIAL: NCT07023120
Title: Optimizing PENG Block in Hip Arthroplasty: Influence of Ropivacaine Volume and Dexamethasone on Analgesic Efficacy
Brief Title: PENG Block Optimization: Volume and Dexamethasone Effects
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8/2025
Record Dates: First submitted 2025-06-08; First posted 2025-06-15 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-06

CONDITIONS: Hip Arthropathy; Hip Osteoarthritis; Hip Arthritis
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Ropivacaine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- PENG 20 mL (Active Comparator): Ultrasound-guided PENG block - 20ml 0,2% ropivacaine
  Interventions: Drug: Ropivacaine 0.2% Injectable Solution
- PENG 20 mL + DEX (Active Comparator): Ultrasound-guided PENG block - 20ml 0,2% ropivacaine + 4mg Dexamethasone
  Interventions: Drug: Ropivacaine 0.2% Injectable Solution; Drug: Dexamethasone 4mg
- PENG 10 mL (Active Comparator): Ultrasound-guided PENG block - 10ml 0,2% ropivacaine
  Interventions: Drug: Ropivacaine 0.2% Injectable Solution
- PENG 10 mL + DEX (Active Comparator): Ultrasound-guided PENG block - 10ml 0,2% ropivacaine + 4mg Dexamethasone
  Interventions: Drug: Dexamethasone 4mg; Drug: Ropivacaine 0.2% Injectable Solution

INTERVENTIONS:
Drug: Ropivacaine 0.2% Injectable Solution — 20ml 0.2% Ropivacaine
  Arms: PENG 20 mL; PENG 20 mL + DEX
Drug: Dexamethasone 4mg — perineural 4mg Dexamethasone
  Arms: PENG 10 mL + DEX; PENG 20 mL + DEX
Drug: Ropivacaine 0.2% Injectable Solution — 10ml 0.2% Ropivacaine
  Arms: PENG 10 mL; PENG 10 mL + DEX

SUMMARY:
This randomized controlled trial investigates the impact of local anesthetic volume and perineural dexamethasone on the analgesic and anti-inflammatory effectiveness of the pericapsular nerve group (PENG) block in patients undergoing total hip arthroplasty (THA). Patients were randomized to receive one of four PENG block variants differing in ropivacaine volume (10 mL or 20 mL of 0.2%) and the addition of 4 mg of perineural dexamethasone. The study evaluates postoperative pain, opioid requirements, systemic inflammatory markers, and quadriceps motor preservation.

DETAILED DESCRIPTION:
The pericapsular nerve group (PENG) block has become a widely used motor-sparing component of multimodal analgesia for total hip arthroplasty (THA). However, its optimal formulation-particularly the volume of local anesthetic and the role of adjuvants-remains undetermined. This prospective, double-blind, randomized controlled trial evaluates the influence of ropivacaine volume (10 mL vs. 20 mL of 0.2%) and the addition of perineural dexamethasone (4 mg) on analgesic efficacy, opioid consumption, systemic inflammation, and quadriceps strength preservation.

A total of 120 adult patients undergoing unilateral THA under spinal anesthesia were randomized to one of four PENG block groups:

Group 1: 20 mL of 0.2% ropivacaine (standard-volume PENG) Group 2: 20 mL of 0.2% ropivacaine + 4 mg perineural dexamethasone Group 3: 10 mL of 0.2% ropivacaine (low-volume PENG) Group 4: 10 mL of 0.2% ropivacaine + 4 mg perineural dexamethasone The primary outcome was the time to first rescue opioid analgesia. Secondary outcomes included total 48-hour opioid consumption (expressed in oral morphine equivalents), numeric rating scale (NRS) pain scores, quadriceps muscle strength, neutrophil-to-lymphocyte ratio (NLR), and platelet-to-lymphocyte ratio (PLR) at 12, 24, and 48 hours postoperatively.

Results demonstrated that the addition of dexamethasone, regardless of volume, significantly prolonged the duration of analgesia and reduced opioid consumption compared to non-adjuvanted PENG blocks. The low-volume + dexamethasone group achieved comparable analgesia to high-volume protocols with better inflammatory profiles. Quadriceps strength was preserved in all groups. These findings support the use of perineural dexamethasone as an effective enhancer of PENG block analgesia while enabling lower local anesthetic volume, potentially improving safety and recovery outcomes in THA patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years scheduled for primary unilateral total hip arthroplasty (THA).
* American Society of Anesthesiologists (ASA) physical status I-III.
* Ability to provide written informed consent.
* Spinal anesthesia planned as the primary anesthetic technique.
* Body mass index (BMI) between 18 and 35 kg/m².
* Fluent in the local language and able to understand the NRS pain scoring system.

Exclusion Criteria:

* Known allergy or hypersensitivity to ropivacaine, dexamethasone, or other amide local anesthetics.
* Pre-existing neurological deficits or neuropathies affecting lower limb motor or sensory function.
* Chronic opioid use (daily use >30 mg oral morphine equivalents for >1 month prior to surgery).
* History of coagulopathy, current anticoagulant therapy not eligible for regional anesthesia.
* Uncontrolled diabetes mellitus (HbA1c > 9%) or active systemic infection.
* Pregnancy or breastfeeding.
* Previous surgery or implantation on the ipsilateral hip.
* Inability to cooperate with postoperative assessments or participate in follow-up.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Time to first rescue opioid | 24 hours after surgery
  Time after surgery when the patient needs opiate for the first time

SECONDARY OUTCOMES:
Total 48h opioid consumption | 48 hours after surgery
  Total opiate consumption after surgery
Numerical Rating Scale [range 0:10] | 4 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Numerical Rating Scale [range 0:10] | 8 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Numerical Rating Scale [range 0:10] | 12 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Numerical Rating Scale [range 0:10] | 24 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Numerical Rating Scale [range 0:10] | 48 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
NLR | 12 hours after surgery
  neutrophile-to-lymphocyte ratio
NLR | 24 hours after surgery
  neutrophile-to-lymphocyte ratio
NLR | 48 hours after surgery
  neutrophile-to-lymphocyte ratio
PLR | 12 hours after surgery
  platelet-to-lymphocyte ratio
PLR | 24 hours after surgery
  platelet-to-lymphocyte ratio
PLR | 48 hours after surgery
  platelet-to-lymphocyte ratio
Quadriceps strength | 4 hours after surgery
  Quadriceps muscle strength (knee extension and hip adduction) will be evaluated according to the medical research council muscle strength rating
Quadriceps strength | 8 hours after surgery
  Quadriceps muscle strength (knee extension and hip adduction) will be evaluated according to the medical research council muscle strength rating
Quadriceps strength | 12 hours after surgery
  Quadriceps muscle strength (knee extension and hip adduction) will be evaluated according to the medical research council muscle strength rating
Quadriceps strength | 24 hours after surgery
  Quadriceps muscle strength (knee extension and hip adduction) will be evaluated according to the medical research council muscle strength rating
Quadriceps strength | 48 hours after surgery
  Quadriceps muscle strength (knee extension and hip adduction) will be evaluated according to the medical research council muscle strength rating
blood glucose | 12 hours after surgery
  blood glucose level
blood glucose | 24 hours after surgery
  blood glucose level
blood glucose | 48 hours after surgery
  blood glucose level
Nerve damage | 12 hours after surgery
  Nerve damage assesment will be performed using the nerve damage score (N0- no nerve damage; N1- minor - sensory paresthesia; N2- major -complete sensory anesthesia; N3- Complete- complete motor defect with or without paraesthesia; N4-CRPS- Complex Regional Pain Syndrome)
Nerve damage | 24 hours after surgery
  Nerve damage assesment will be performed using the nerve damage score (N0- no nerve damage; N1- minor - sensory paresthesia; N2- major -complete sensory anesthesia; N3- Complete- complete motor defect with or without paraesthesia; N4-CRPS- Complex Regional Pain Syndrome)
Nerve damage | 48 hours after surgery
  Nerve damage assesment will be performed using the nerve damage score (N0- no nerve damage; N1- minor - sensory paresthesia; N2- major -complete sensory anesthesia; N3- Complete- complete motor defect with or without paraesthesia; N4-CRPS- Complex Regional Pain Syndrome)

CONTACTS AND LOCATIONS:
Overall Officials: Malgorzata Reysner, M.D. Ph.D., Study Chair — Poznan University of Medical Sciences
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No